CLINICAL TRIAL: NCT03603158
Title: Influence of KCNH2 Polymorphisms on the QTc Interval in Kelantanese Malays Patients Receiving Methadone Maintenance Therapy (MMT) in Malaysia
Brief Title: KCNH2 Polymorphisms on the QTc Interval in Kelantanese Malays Patients Receiving Methadone Maintenance Therapy (MMT)
Status: Completed | Type: Observational
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Muhammad Irfan Abdul Jalal, Principal Investigator, Universiti Sains Malaysia
Other Study IDs: USMKK/PPP/JEPeM 9221.3[5]
Record Dates: First submitted 2018-07-18; First posted 2018-07-27 (Actual); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: Opioid Dependence; Methadone Toxicity; HERG Gene Mutation
Keywords: HERG; KCNH2; METHADONE; OPIOID
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Genomic DNA extracted from peripheral leukocytes in 5 mls venous blood samples provided by all methadone recipients enrolled in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Methadone maintenance therapy (MMT) is one of the modalities to prevent HIV transmission among injected drug users, particularly in opioid-dependent users. However, methadone-associated cardiotoxicity is one of the fatal adverse events that limit the widespread usage in certain groups of opioid-dependent patients. This is a cross-sectional study aimed to investigate the association between 4 KCNH2 SNPs (1539C>T, in exon 6 of KCNH2 gene; 1956T>C, in exon 8 of KCNH2 gene), 2350C>T (in exon 9 of KCNH2 gene), 2690A>C (Exon 11 of KCNH2 gene)) and prolongation of QTc interval in opioid-dependent Kelantanese Malays who are the recipients of Methadone Maintenance Therapy. The investigators hypothesized that subjects with minor alleles of those 4 SNPs will have longer QTc intervals than those with major alleles, adjusting for the effects of other confounding factors such as age and gender of the subjects, plasma methadone trough levels, hypokalemia, hypocalcemia and hypomagnesemia. The investigators also aimed to provide a model that will reliably predict the magnitude QTc based on the SNPs data and other covariates mentioned above. This will greatly assist in identifying methadone recipients who are at risk of developing prolonged QTc or the more fatal torsade de pointes.

DETAILED DESCRIPTION:
Introduction

Methadone maintenance therapy (MMT) is one of the modalities to prevent HIV transmission among injected drug users, particularly in opioid-dependent users. However, methadone-associated cardiotoxicity is one of the fatal adverse events that limit the widespread usage in certain groups of opioid-dependent patients.

Study hypotheses / aims

The investigators hypothesized that subjects with minor alleles of those 4 SNPs would have longer QTc intervals than those with major alleles, adjusting for the effects of other confounding factors such as age and gender of the subjects, plasma methadone trough levels, hypokalemia, hypocalcemia and hypomagnesemia. The investigators also aimed to provide a model that will reliably predict the magnitude QTc based on the SNPs data and other covariates mentioned above. This will greatly assist in identifying methadone recipients who are at risk of developing prolonged QTc or the more fatal torsade de pointes.

Study Design and Sample Size Calculation

This is a cross-sectional study aimed to investigate the association between 4 KCNH2 SNPs (1539C>T, in exon 6 of KCNH2 gene; 1956T>C, in exon 8 of KCNH2 gene), 2350C>T (in exon 9 of KCNH2 gene), 2690A>C (Exon 11 of KCNH2 gene)) and prolongation of QTc interval in opioid-dependent Kelantanese Malays who are the recipients of Methadone Maintenance Therapy . The sample size was calculated using single-proportion formula and the information required was based on a similar prior study conducted among Singaporean Malay. It was concluded that the sample size required is 105 patients. Since eligible patients were lacking, the convenience (non-probability) sampling method was used.

During the initial visit, relevant clinico-demographic details such as age, gender, history of drug addiction and psychiatric illnesses, drug dependency patterns, other drug usage and treatment-related issues for each patient were gathered. Subsequently a validated Malay version of Subjective Opioid Withdrawal Scale (SOWS) questionnaire was administered to assess any opioid withdrawal symptoms experienced by study participants.

Five (5) mls of blood was then withdrawn for each subject for the ascertainment of relevant biochemical profile (serum potassium, magnesium, calcium), plasma methadone trough levels, and KCNH2 SNPs genotyping. Drug screening for substances such as MDMA, benzodiazepines methamphetamine, cannabis, marijuana were also carried out using urine dipstick test at urine collection point. The colour and temperature of the urine were also recorded.

QT measurement was obtained using calibrated Welch Allyn CP 50™ ECG (Electrocardiograph) (Welch Allyn Australia Pty Ltd., New South Wales, Australia) machine, printed at a paper speed of 25mm/s and voltage of 10mm/mV. QTc measurement was then manually calculated using Fredericia's formula to correct for heart rate (R-R interval). All trained personnel who were responsible for obtaining QTc measurement from each patient were blinded to other information on serum biochemical profiles and methadone trough levels.

KCNH2 Genotyping

The DNA was extracted according to procedures modified from Bethesda Research Laboratories based on the revisions made to the Brinboam and Doly method. The quantity and quality of the extracted DNA were determined using NanoDrop ND-1000 Spectrophotometer (NanoDrop Technologies, Inc. Wilmington, USA) with measurements done at 260 and 280 nm. The integrity of the extracted DNA was determined using 2% agarose gel electrophoresis performed at 70 Volts for 90 minutes.

The DNA in all samples were amplified for all 4KCNH2 SNPs were performed using 2-step nested allele-specific multiplex polymerase chain reaction (PCR). The primers (both forward and reverse) were designed according to the published sequence for KCNH2 (NC_000007.13). To improve primer specificity, mismatch at its 3´ ends that were specific to either the variant sequence or wild-type DNA sequence at the specified locus was made to the primers. Besides, the primers were also designed and manipulated to differentiate between the different single nucleotide changes/alleles during PCR amplification. To verify primers specificity, the BLAST program at NCBI (http://www.ncbi.nlm.nih.gov/ blast) was used.

In the first multiplex PCR, exon 6,8,9 and 11 were amplified under the following condition: pre-denaturation at 95°C for 1 minute followed by 25-cycle of denaturation at 95°C for 15 seconds, annealing for 65°C for 15 seconds, and extension at 72°C for 10 seconds. Upon full 25-cycle completion, final extension phase lasted for 72°C for 7 minutes. The PCR products (amplicons) were then resolved using 2% agarose gel electrophoresis at 130 Volts for 90 minutes.

The PCR products of the first multiplex PCR were then used as templates for second PCR which targeted the 4 respective SNPs region for amplification. This was performed under the following condition:pre-denaturation at 95°C for 1 minute followed by 25-cycle of denaturation at 95°C for 15 seconds, annealing for 69°C for 30 seconds, and extension at 72°C for 4 seconds. Upon full 25-cycle completion, final extension phase lasted for 72°C for 7 minutes. The PCR products (amplicons) were then resolved using 2% agarose gel electrophoresis at 130 Volts for 90 minutes.

The first products of the amplified regions in the Exons 6, 8, 9, and Exon11 were subsequently submitted for direct DNA sequencing. QIAquick PCR purification kit (Qiagen, USA) was used for purification of the PCR products. DNA sequencing was carried out by applying 3130XL genetic analyzer DNA sequencer (ABI, USA). The results were compared with the published sequences for KCNH2 in the NCBI, accession number (NC_000007.13)

Statistical Analysis

The select equally likely or more extreme samples (SELOME) version of the Fisher's exact test was employed to examine whether the distribution of the SNP alleles and genotype follow the Hardy-Weinberg Equilibrium (HWE) assumption. Those SNPs that significantly deviated from the HWE assumption were dropped from further analysis.

To examine the associations between the 4SNPs and QTc interval (measured as continuous variable) and build a statistical model that can reliably predict QTc intervals, simple and multiple linear regression methods were used. Age and gender of the patients, plasma methadone trough levels, serum potassium, calcium and magnesium were treated as confounding factors whose effects on QTc were adjusted for.

ELIGIBILITY:
Inclusion Criteria:

* Opioid-dependent subjects aged 18 years and above
* Opioid-dependent subjects who were on Methadone Maintenance Therapy (MMT) for 6 months or longer and had stable plasma methadone concentration
* Malay ancestry up to 3 generations
* A history of good compliance with Directly-Observed Therapy (DOT)

Exclusion Criteria:

* Opioid-dependent subjects who were aggressive and had active psychiatric illnesses
* Opioid-dependent subjects with chronic medical and surgical illnesses
* Opioid-dependent subjects with cardiac structural defects
* Inability to communicate in Malay or English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Kelantanese Malay opioid-dependent subjects who were on Methadone Maintenance Therapy (MMT) in the Eastern-coastal state of Kelantan, Malaysia.
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2011-02-01 (Actual); Primary Completion 2012-12-31 (Actual); Study Completion 2012-12-31 (Actual)

PRIMARY OUTCOMES:
QTc Interval | First screening visit
  QT interval (measured in milliseconds) obtained from ECG reading that is then divided by the shortest R-R interval to the power of 0.33 (Fredericia's formula).

CONTACTS AND LOCATIONS:
Overall Officials: Muslih AbdulKarim Ibrahim, PhD, Principal Investigator — Hawler University
Locations (1):
- Hospital Universiti Sains Malaysia, Kubang Kerian, Kelantan, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Koo SH, Ho WF, Lee EJ. Genetic polymorphisms in KCNQ1, HERG, KCNE1 and KCNE2 genes in the Chinese, Malay and Indian populations of Singapore. Br J Clin Pharmacol. 2006 Mar;61(3):301-8. doi: 10.1111/j.1365-2125.2005.02545.x. PMID 16487223
- [Result] Hajj A, Ksouda K, Peoc'h K, Curis E, Messali A, Deveaux LL, Bloch V, Prince N, Mouly S, Scherrmann JM, Lepine JP, Laplanche JL, Drici MD, Vorspan F. KCNH2 polymorphism and methadone dosage interact to enhance QT duration. Drug Alcohol Depend. 2014 Aug 1;141:34-8. doi: 10.1016/j.drugalcdep.2014.04.027. Epub 2014 May 14. PMID 24875677
- See also: Abstract and full text — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC1885019/
- See also: Abstract — https://www.ncbi.nlm.nih.gov/pubmed/24875677